CLINICAL TRIAL: NCT03612336
Title: Substudy of Efficacy, Safety and Toxicology of Electronic Nicotine Delivery Systems as an Aid for Smoking Cessation (ESTxENDS Trial)- the Metabolic Substudy of ESTxENDS
Brief Title: The ESTxENDS Trial- Substudy on the Metabolic Effects of Using Electronic Nicotine Delivery Systems (ENDS/Vaporizer/E-cig)
Acronym: ESTxENDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bern (Other)
Collaborators: University of Lausanne (Other); University of Geneva, Switzerland (Other); University of Zurich (Other); State Hospital, St. Gallen (Other Government); Swiss National Science Foundation (Other); Krebsforschung Schweiz, Bern, Switzerland (Other); Federal Office of Public Health, Switzerland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2017-02332b
Record Dates: First submitted 2018-06-25; First posted 2018-08-02 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-11

CONDITIONS: Smoking Cessation; Cardiovascular Diseases
MeSH Terms: conditions — Smoking Cessation; Cardiovascular Diseases

STUDY DESIGN:
Masking Description: Statisticians and laboratory personnel will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Other: ENDS (vaporizer/e-cig) and smoking cessation counseling
- Control group (Active Comparator)
  Interventions: Other: Smoking cessation counseling

INTERVENTIONS:
Other: ENDS (vaporizer/e-cig) and smoking cessation counseling — Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Intervention group
Other: Smoking cessation counseling — Participants in the control group will receive smoking cessation counseling only. Participants will be allowed to additionally use nicotine replacement therapy. All participants will be followed over a 24-month period. Smoking cessation counseling will be provided in person at the first clinical visit and then over the phone at the target quit date one week later and again at week 2, 4 and 8 after the target quit date. After 6, 12 and 24 months, participants will be asked to come to a clinical visit.
  Arms: Control group

SUMMARY:
--> This is a substudy of the main ESTxENDS trial (NCT03589989). Metabolic outcomes should be considered secondary outcomes of the main smoking cessation outcome formulated in NCT03589989.

Cardiovascular diseases (CVD) are a leading cause of death in cigarette smokers; quitting smoking is associated with reduced CVD. Cigarette smoking increases CVD through complex mechanisms, mostly on an increase in atherosclerosis and the effect appears unrelated to nicotine. Recently, electronic nicotine delivery systems (ENDS; also called vaporizer or electronic cigarette) have become popular with smokers who want to stop smoking. There is currently no evidence that ENDS use affects CVD outcomes. The nicotine contained in the e-liquids from ENDS has cardiovascular effects and the evidence about health effects mostly comes from studies on nicotine replacement therapy (NRT). These studies did not show an increased risk of CVD from NRTs. The ECLAT trial showed no difference in body weight, resting heart rate, or blood pressure between those who used ENDS or not. Two studies evaluated the short-term effects of ENDS on the cardiovascular system. One study suggested impairment in diastolic ventricular function with cigarettes and not with ENDS. Both ENDS and cigarettes increased diastolic blood pressure, potentially mediated through nicotine exposure, but an increased systolic blood pressure was found only in cigarette smokers. Other studies have suggested no changes in blood pressure in daily users of electronic cigarettes up to 1 year with some even a reduction in blood pressure among patients with hypertension. Interventions helping smokers quit have shown that quitting is associated with increased HDL-cholesterol, weight gain, higher blood glucose, and higher diabetes risk. No large randomized trials have tested the effect of ENDS on blood cholesterol and other markers of cardiovascular risk.

This study will therefore test the efficacy of ENDS for cigarette smoking cessation, the safety of ENDS on adverse events and the effect of ENDS on health-related outcomes and exposure to inhaled chemicals.

For the main ESTxENDS trial (NCT03589989), smokers motivated to quit smoking cigarettes will be included. Participants in the intervention group will receive an ENDS and nicotine-containing e-liquids, which they will be allowed to use ad libitum. Additionally, they will receive smoking cessation counseling. Participants in the control group will receive smoking cessation counseling only. All participants will be followed over a 24-month period. Measurements of risk factors for cardiovascular diseases will be done at baseline and at 6, 12 and 24 months' follow-up.

ELIGIBILITY:
Inclusion criteria:

* Informed Consent as documented by signature
* Persons aged 18 or older
* Currently smoking 5 or more cigarettes a day for at least 12 months
* Willing to try to quit smoking within the next 3 months,
* Persons providing a valid phone number, a valid email address and/or a valid postal address.

Exclusion criteria:

* Known hypersensitivity or allergy to contents of the e-liquid
* Participation in another study with investigational drug within the 30 days preceding the baseline visit and during the present study where interactions are to be expected
* Women who are pregnant or breast feeding
* Intention to become pregnant during the course of the scheduled study intervention, i.e. within the first 6-months of the study
* Persons having used ENDS or tobacco heating systems regularly in the 3 months preceding the baseline visit
* Persons having used nicotine replacement therapy (NRT) or other medications with demonstrated efficacy as an aid for smoking cessation such as varenicline or bupropion within the 3 months preceding the baseline visit
* Persons who cannot attend the 6- month follow-up visit for any reason
* Cannot understand instructions delivered in person or by phone, or otherwise unable to participate in study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1246 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Measurements of risk factors for cardiovascular diseases (blood pressure)_1 | 6 months post quit date
  Measurement of blood pressure
Measurements of risk factors for cardiovascular diseases (blood pressure)_2 | 12 months post quit date
  Measurement of blood pressure
Measurements of risk factors for cardiovascular diseases (blood pressure)_3 | 24 months post quit date
  Measurement of blood pressure
Measurements of risk factors for cardiovascular diseases (heart rate)_1 | 6 months post quit date
  Measurement of heart rate
Measurements of risk factors for cardiovascular diseases (heart rate)_2 | 12 months post quit date
  Measurement of heart rate
Measurements of risk factors for cardiovascular diseases (heart rate)_3 | 24 months post quit date
  Measurement of heart rate
Measurements of risk factors for cardiovascular diseases (total cholesterol)_1 | 6 months post quit date
  Measurement of total cholesterol
Measurements of risk factors for cardiovascular diseases (total cholesterol)_2 | 12 months post quit date
  Measurement of total cholesterol
Measurements of risk factors for cardiovascular diseases (total cholesterol)_3 | 24 months post quit date
  Measurement of total cholesterol
Measurements of risk factors for cardiovascular diseases (LDL-cholesterol)_1 | 6 months post quit date
  Measurement of LDL-cholesterol
Measurements of risk factors for cardiovascular diseases (LDL-cholesterol)_2 | 12 months post quit date
  Measurement of LDL-cholesterol
Measurements of risk factors for cardiovascular diseases (LDL-cholesterol)_3 | 24 months post quit date
  Measurement of LDL-cholesterol
Measurements of risk factors for cardiovascular diseases (HDL-cholesterol)_1 | 6 months post quit date
  Measurement of HDL-cholesterol
Measurements of risk factors for cardiovascular diseases (HDL-cholesterol)_2 | 12 months post quit date
  Measurement of HDL-cholesterol
Measurements of risk factors for cardiovascular diseases (HDL-cholesterol)_3 | 24 months post quit date
  Measurement of HDL-cholesterol
Measurements of risk factors for cardiovascular diseases (triglycerides)_1 | 6 months post quit date
  Measurement of triglycerides
Measurements of risk factors for cardiovascular diseases (triglycerides)_2 | 12 months post quit date
  Measurement of triglycerides
Measurements of risk factors for cardiovascular diseases (triglycerides)_3 | 24 months post quit date
  Measurement of triglycerides
Measurements of risk factors for cardiovascular diseases (HbA1c)_1 | 6 months post quit date
  Measurement of HbA1c for persons with diagnosed diabetes
Measurements of risk factors for cardiovascular diseases (HbA1c)_2 | 12 months post quit date
  Measurement of HbA1c for persons with diagnosed diabetes
Measurements of risk factors for cardiovascular diseases (HbA1c)_3 | 24 months post quit date
  Measurement of HbA1c for persons with diagnosed diabetes
Measurements of risk factors for cardiovascular diseases (creatinine)_1 | 6 months post quit date
  Measurement of creatinine
Measurements of risk factors for cardiovascular diseases (creatinine)_2 | 12 months post quit date
  Measurement of creatinine
Measurements of risk factors for cardiovascular diseases (creatinine)_3 | 24 months post quit date
  Measurement of creatinine
Measurements of risk factors for cardiovascular diseases (waist circumference)_1 | 6 months post quit date
  Measurement of waist circumference
Measurements of risk factors for cardiovascular diseases (waist circumference)_2 | 12 months post quit date
  Measurement of waist circumference
Measurements of risk factors for cardiovascular diseases (waist circumference)_3 | 24 months post quit date
  Measurement of waist circumference
Measurements of risk factors for cardiovascular diseases (body mass index, BMI)_1 | 6 months post quit date
  Measurements of weight and height to report BMI in kg/m^2
Measurements of risk factors for cardiovascular diseases (body mass index, BMI)_2 | 12 months post quit date
  Measurements of weight and height to report BMI in kg/m^2
Measurements of risk factors for cardiovascular diseases (body mass index, BMI)_3 | 24 months post quit date
  Measurements of weight and height to report BMI in kg/m^2

SECONDARY OUTCOMES:
Changes in cardiovascular disease risk factors (blood pressure) | Change from Baseline to 6,12, 24 months post quit date
  Measurement of blood pressure
Changes in cardiovascular disease risk factors (heart rate) | Change from Baseline to 6,12, 24 months post quit date
  Measurement of heart rate
Changes in cardiovascular disease risk factors (total cholesterol) | Change from Baseline to 6,12, 24 months post quit date
  Measurement of total cholesterol
Changes in cardiovascular disease risk factors (LDL-cholesterol) | Change from Baseline to 6,12, 24 months post quit date
  Measurement of LDL-cholesterol
Changes in cardiovascular disease risk factors (HDL- cholesterol) | Change from Baseline to 6,12, 24 months post quit date
  Measurement of HDL- cholesterol
Changes in cardiovascular disease risk factors (triglycerides) | Change from Baseline to 6,12, 24 months post quit date
  Measurement of triglycerides
Changes in cardiovascular disease risk factors (HbA1c) | Change from Baseline to 6,12, 24 months post quit date
  Measurement of HbA1c for persons with diagnosed diabetes
Changes in cardiovascular disease risk factors (creatinine) | Change from Baseline to 6,12, 24 months post quit date
  Measurement of creatinine
Changes in cardiovascular disease risk factors (waist circumference) | Change from Baseline to 6,12, 24 months post quit date
  Measurement of waist circumference
Changes in cardiovascular disease risk factors (body mass index, BMI) | Change from Baseline to 6,12, 24 months post quit date
  Measurements of weight and height to report BMI in kg/m^2
Physical activity | 6,12, 24 months post quit date
  Measured using the International Physical activity questionnaire (IPAQ). The short version (7 items) provides information on the time spent walking, in vigorous- and moderate-intensity activity and in sedentary activity.
Changes of physical activity | Change from Baseline to 6,12, 24 months post quit date
  Measured using the International Physical activity questionnaire (IPAQ). The short version (7 items) provides information on the time spent walking, in vigorous- and moderate-intensity activity and in sedentary activity.

CONTACTS AND LOCATIONS:
Overall Officials: Reto Auer, Prof.Dr.med, Study Director — Berner Institut für Hausarztmedizin; Universität Bern
Locations (5):
- Switzerland (5):
  - Unisanté, Centre universitaire de médecine générale et santé publique, Université de Lausanne, Lausanne, Canton of Vaud
  - University Clinic for General Internal Medicine, Bern University Hospital, Bern
  - Département de médecine interne, Hôpitaux universitaires de Genève, Geneva
  - Lungenzentrum, Klinik für Pneumologie und Schlafmedizin, Kantonsspital St. Gallen, Sankt Gallen
  - Epidemiology, Biostatistics and Prevention Institute (EBPI), University of Zurich, Zurich

REFERENCES:
- [Background] Jha P, Ramasundarahettige C, Landsman V, Rostron B, Thun M, Anderson RN, McAfee T, Peto R. 21st-century hazards of smoking and benefits of cessation in the United States. N Engl J Med. 2013 Jan 24;368(4):341-50. doi: 10.1056/NEJMsa1211128. PMID 23343063
- [Background] Benowitz NL, Pipe A, West R, Hays JT, Tonstad S, McRae T, Lawrence D, St Aubin L, Anthenelli RM. Cardiovascular Safety of Varenicline, Bupropion, and Nicotine Patch in Smokers: A Randomized Clinical Trial. JAMA Intern Med. 2018 May 1;178(5):622-631. doi: 10.1001/jamainternmed.2018.0397. PMID 29630702
- [Background] Benowitz NL, Fraiman JB. Cardiovascular effects of electronic cigarettes. Nat Rev Cardiol. 2017 Aug;14(8):447-456. doi: 10.1038/nrcardio.2017.36. Epub 2017 Mar 23. PMID 28332500
- [Background] Caponnetto P, Campagna D, Cibella F, Morjaria JB, Caruso M, Russo C, Polosa R. EffiCiency and Safety of an eLectronic cigAreTte (ECLAT) as tobacco cigarettes substitute: a prospective 12-month randomized control design study. PLoS One. 2013 Jun 24;8(6):e66317. doi: 10.1371/journal.pone.0066317. Print 2013. PMID 23826093
- [Background] Farsalinos KE, Tsiapras D, Kyrzopoulos S, Savvopoulou M, Voudris V. Acute effects of using an electronic nicotine-delivery device (electronic cigarette) on myocardial function: comparison with the effects of regular cigarettes. BMC Cardiovasc Disord. 2014 Jun 23;14:78. doi: 10.1186/1471-2261-14-78. PMID 24958250
- [Background] Farsalinos K, Cibella F, Caponnetto P, Campagna D, Morjaria JB, Battaglia E, Caruso M, Russo C, Polosa R. Effect of continuous smoking reduction and abstinence on blood pressure and heart rate in smokers switching to electronic cigarettes. Intern Emerg Med. 2016 Feb;11(1):85-94. doi: 10.1007/s11739-015-1361-y. Epub 2016 Jan 9. PMID 26749533
- [Background] Oncken CA, Litt MD, McLaughlin LD, Burki NA. Nicotine concentrations with electronic cigarette use: effects of sex and flavor. Nicotine Tob Res. 2015 Apr;17(4):473-8. doi: 10.1093/ntr/ntu232. PMID 25762758
- [Background] Forey BA, Fry JS, Lee PN, Thornton AJ, Coombs KJ. The effect of quitting smoking on HDL-cholesterol - a review based on within-subject changes. Biomark Res. 2013 Sep 13;1(1):26. doi: 10.1186/2050-7771-1-26. PMID 24252691
- [Background] Aubin HJ, Farley A, Lycett D, Lahmek P, Aveyard P. Weight gain in smokers after quitting cigarettes: meta-analysis. BMJ. 2012 Jul 10;345:e4439. doi: 10.1136/bmj.e4439. PMID 22782848
- [Background] Stein JH, Asthana A, Smith SS, Piper ME, Loh WY, Fiore MC, Baker TB. Smoking cessation and the risk of diabetes mellitus and impaired fasting glucose: three-year outcomes after a quit attempt. PLoS One. 2014 Jun 3;9(6):e98278. doi: 10.1371/journal.pone.0098278. eCollection 2014. PMID 24893290